CLINICAL TRIAL: NCT06099665
Title: Addressing Under-treatment and Health Equity in Aortic Stenosis and Mitral Regurgitation Using an Integrated EHR Platform
Brief Title: Addressing Under-treatment and Health Equity in AS and MR Using an Integrated EHR Platform
Acronym: ALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tempus AI (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TMPS-Cardio-01
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Aortic Valve Stenosis; Mitral Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated alert (Experimental): Providers that will receive an automated alert sent via the EHR.
  Interventions: Behavioral: Automated alert
- Control (No Intervention): Care providers in the control arm will not receive an automated alert.

INTERVENTIONS:
Behavioral: Automated alert — Receiving an automated alert via the EHR to highlight that the patient in question presents for severe aortic stenosis or severe mitral regurgitation according to the AHA guidelines and that they are a good candidate for valve intervention. The alert will not list any specific manufacturer's device.
  Arms: Automated alert

SUMMARY:
This multi-center, prospective, cluster-randomized controlled trial will evaluate Tempus Next automated notifications as an intervention to support identification and evaluation of patients possibly indicated for Valve Intervention (VI). This study will evaluate the impact of Tempus Next's automated notifications on: (1) Transcatheter or surgical procedure for AS or MR; and (2) Clinic visit with at least one member of the Multidisciplinary Heart Team (including time to evaluation) for patients with definitive or possible severe AS or MR on echocardiogram. These endpoints will also be examined within and between assigned groups according to race, ethnicity, sex, and geography.

The primary question that will be answered:

Do automated alerts sent to clinical providers decrease under-treatment of severe aortic stenosis and severe mitral regurgitation?

The study will compare the rate of clinical follow-up and aortic valve surgery in a control group (no alerts sent) to a treatment group (alerts sent to an appropriate care provider).

ELIGIBILITY:
At least one of the following three options for aortic stenosis and/or the single option for mitral regurgitation are determined from echocardiogram findings:

1. AVA or DI (Patients with either Aortic valve area (AVA) or Dimensionless Index (DI) measured in their echo as well as at least one hemodynamic measure above the minimum threshold)

   a. Either: i. Aortic Valve Area ≤ 1.0 cm2 ii. Dimensionless Index ≤ 0.25 b. AND ANY of i. Aortic Mean Gradient ≥ 15 mmHg ii. Aortic Peak Gradient ≥ 30 mmHg iii. Aortic Jet Velocity ≥ 2.75 m/s
2. AVA + OTHER (Patients with AVA and at least 1 other echo measurement in their echo above the threshold)

   1. 1.0 cm2 < Aortic Valve Area ≤ 1.2 cm2
   2. AND ANY of:

   i. Aortic Mean Gradient ≥ 40 mmHg ii. Aortic Peak Gradient ≥ 64 mmHg iii. Aortic Jet Velocity ≥ 4.0 m/s
3. POSSIBLE (Possible Aortic Stenosis but requires human review) a. Aortic Valve Area is NULL OR >1.2 cm2 b. AND ANY of: i. Aortic Mean Gradient ≥ 40 mmHg ii. Aortic Peak Gradient ≥ 64 mmHg iii. Aortic Jet Velocity ≥ 4.0 m/s OR a. EITHER i. Aortic Valve Area ≤ 1.0 cm2 ii. Dimensionless Index ≤ 0.25 b. AND ALL are: i. Aortic Mean Gradient < 15 mmHg ii. Aortic Peak Gradient < 30 mmHg iii. Aortic Peak Velocity < 2.75 m/s

ALERT Study Clinical Investigation Plan Version 2.1 page 12 of 54

Any patient flagged for "POSSIBLE" does not result in automatically alerting the provider, instead a notification is sent to the Tempus research team for manual review in conjunction with the site Principal Investigator (PI) and if requested by Tempus or site PI, a Steering Committee member. If clinical confirmation is received for severe aortic stenosis from the site PI, an alert is sent to the provider. 1. Mitral Regurgitation

a. Mention of severe mitral regurgitation or moderate- severe mitral regurgitation

Any patient mentioned with only moderate MR or a lesser severity will be excluded.

Exclusion Criteria:

1. Age < 18 years
2. Patient had evidence of a prior transcatheter or surgical repair or replacement of the target valve
3. The echocardiogram was ordered by a cardiologist on the MHT or a cardiac surgeon
4. Patient already has a scheduled clinic visit with a member of the MHT or a recent (since the start of the study at that site ) clinic visit with the MHT, or a scheduled transcatheter or surgical VI in the future.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2626 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Establish impact of automated alerts on the hierarchical composite endpoint of valve intervention (VI) or follow-up visit with a multi-disciplinary heart team (MHT). | 90 days from a qualifying echocardiogram indicating severe aortic stenosis or mitral regurgitation
  Determining whether an automated alert improves recognition and management of severe AS and severe MR through its impact on the utilization of VI or follow-up visit with MHT, which is defined as the proportion of patients with a clinical indication for severe AS or severe MR that undergo VI or have a follow-up visit with MHT. We will utilize an automated alert to highlight TTE results that are consistent with or may be consistent with severe AS and severe MR for patients that do not have a scheduled follow-up with the MHT or an AVR procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Batchelor, MD, Principal Investigator — Director of Interventional Cardiology Inova Heart and Vascular Institute
Locations (6):
- United States (6):
  - Saint Luke's Health System, Kansas City, Missouri
  - OhioHealth, Columbus, Ohio
  - Bon Secours Mercy Health - Lima Market, Lima, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt, Nashville, Tennessee
  - Bon Secours Mercy Health - Richmond Market, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No